CLINICAL TRIAL: NCT04787224
Title: Soft and Hard Tissue Evaluation for Vestibular Socket Therapy of Immediately Placed Implants in Infected and Non-infected Sockets: A 1-year Prospective Cohort Study
Brief Title: Vestibular Socket Therapy (VST) in Infected and Non Infected Sockets
Acronym: VST
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Collaborators: BioHorizons, Inc. (Industry)
Responsible Party: Principal Investigator, Iman Abd-ElWahab Radi, PhD, Professor, Cairo University
Other Study IDs: 0010557
Record Dates: First submitted 2021-03-04; First posted 2021-03-08 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Implant Site Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- infected sockets: Signs of infection were periapical radiolucency only in 3 sites (2 patients), fistula in 2 sites (2 patients), sinus in 11 sites (7 patients) and finally swelling in 3 sites (2 patients)
  Interventions: Other: immediate implant with vestibular socket therapy
- Non infected sockets: This is ensured by the absence of any clinical signs and symptoms of infection in addition to negative radiographic findings
  Interventions: Other: immediate implant with vestibular socket therapy

INTERVENTIONS:
Other: immediate implant with vestibular socket therapy — A 1-cm long vestibular access incision was cut, 3-4 mm apical to the mucogingival junction of the involved tooth. The socket orifice and the vestibular access incision were connected by a subperiosteal tunnel that was created using a periotome and a micro-periosteal elevator. Implants were installed using a CADLCAM surgical guide. A flexible cortical membrane shield of heterologous origin, 0.6 mm in thickness was prepared by hydrating and trimming it. It was then tucked through the vestibular access incision, till it extended 1 mm below the socket orifice, and stabilized using a membrane tack ( to the apical bone. The gap between the implant and the shield/the labial plate was then filled with particulate bone graft [75% autogenous bone chips harvested form local surgical sites and 25% inorganic bovine bone mineral matrix.
  Other Names: VST

SUMMARY:
Vestibular socket therapy with immediate implant placement is compared in infected and non-infected sockets regarding implant survival, bone thickness and soft tissue height .

DETAILED DESCRIPTION:
For non infected sockets, a 15c blade (Stoma, Storz am Mark GmbH, Emmingen-Liptingen Germany) was used to cut a 1-cm long vestibular access incision , 3-4 mm apical to the mucogingival junction of the involved tooth. The socket orifice and the vestibular access incision were connected by a subperiosteal tunnel that was created using a periotome and a micro-periosteal elevator (Stoma, Storz am Mark GmbH, Emmingen-Liptingen Germany). Implants, (Biohorizons, Birmingham, Al, USA) , were installed using a 3D printed surgical guide (Surgical Guide Resin, Form 2, Formlabs). A flexible cortical membrane shield (OsteoBiol® Lamina, Tecnoss®, Torino, Italy) of heterologous origin, 0.6 mm in thickness was prepared by hydrating and trimming it. It was then tucked through the vestibular access incision, till it extended 1 mm below the socket orifice, and stabilized using a membrane tack (AutoTac System Kit, Biohorizons Implant Systems, Birmingham, Alabama Inc, USA) to the apical bone. The gap between the implant and the shield/the labial plate was then filled with particulate bone graft [75% autogenous bone chips harvested form local surgical sites and 25% inorganic bovine bone mineral matrix (MinerOss X , Biohorizons, Birmingham, Al, USA)]. For the infected sockets, the 6-day protocol was implemented. Atraumatic extraction of the infected tooth by the periotome was followed by curettage, mechanical debridement and chemical irrigation using metronidazole irrigation solution (500mg/100ml, Amrizole, Amria Pharma, Alexandria, Egypt). The root of the involved tooth was cleaned with an ultrasonic cleaner, cut to its apical third, reimplanted into the socket and maintained there for 6 days by bonding its crown to the adjacent teeth using composite resin. Implant and crown placement were done as described above for the non-infected socket group.

ELIGIBILITY:
Inclusion Criteria:

* all patients were adults ≥ 18 years,
* 1-5 non-adjacent hopeless maxillary teeth in the esthetic zone.
* The involved teeth had type II sockets.
* To achieve optimum primary stability for the implants (30Ncm insertion torque), adequate palatal and at least 3 mm apical bone should be available to engage the immediately placed implants.

Exclusion Criteria:

* Smoking and/or pregnant patients
* systemic diseases
* a history of chemo- or radiotherapy within the past 2 years were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with fresh extraction sockets in the esthetic zone
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
implant survival | implant insertion- 1 year
  Implant survival was reported as defined by Buser et al by the absence of peri-implant infection, persistent subjective complaints such as pain, foreign body sensation, and/or dysesthesia, radiolucency around the implant, and/or any detectable implant mobility.

SECONDARY OUTCOMES:
mucosal recession | crown insertion- 1 year
  Amount of mucosal recession was identified midfacially and at the apex of the mesial and distal papillae by superimposing the STL files of the models, obtained via intra-oral scanning, at the baseline (of the unrestorable tooth) with those after 12 months of implant insertion. The 3D software roughly aligned of both pre-and postoperative models through 3 identical points, identified on their surfaces. The best-fit algorithm of the software then perfected the superimposition process. The superimposed models were then imported into an STL viewer, where the measurements were performed. This method was proven to be accurate in volumetric measurements of hard and soft tissues.
labial plate thickness changes | implant insertion- 1 year
  . Changes in the thickness of the labial plate of bone was measured by superimposing CBCT images obtained at the baseline (time of tooth extraction) and those after 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Iman Radi, PhD, Principal Investigator — Cairo University; AbdelSalam Alaskary, BDS, Study Director — Private Practice
Locations (2):
- Egypt (2):
  - Faculty of dentistry, Cairo, Manial
  - ElAskary and Associates Private clinic, Alexandria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elaskary A, Thabet A, Hussin M, Radi IA. Soft and hard tissue evaluation for vestibular socket therapy of immediately placed implants in infected and non-infected sockets: a 1-year prospective cohort study. BMC Oral Health. 2024 Oct 7;24(1):1190. doi: 10.1186/s12903-024-04905-3. PMID 39375634